CLINICAL TRIAL: NCT06113289
Title: A Phase 1B/2A Trial of Combination of ASTX727 With ASTX029 in Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0840; NCI-2023-09243 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-25; First posted 2023-11-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1B (Experimental): During cycle 1: Participants will take: ASTX029 tablets daily by mouth on days 1-42. ASTX727 tablets by mouth 1 time every day on Days 15-19. You should take ASTX727 and ASTX029 fasting (about 2 hours before a meal, and 2 hours after a meal).
  Cycles 2 and beyond: Participants will take ASTX029 tablets by mouth every day (days 1-28) fasting, (2 hours before and 2 hours after a meal). You will also take ASTX727 tablets by mouth 1 time every day on days 1-5 of each cycle, fasting (2 hours before and 2 hours after a meal).
  Interventions: Drug: ASTX727; Drug: ASTX029-01
- Part 2 (Experimental): During cycle 1: Participants will take: ASTX029 tablets daily by mouth on days 1-42. ASTX727 tablets by mouth 1 time every day on Days 15-19. You should take ASTX727 and ASTX029 fasting (about 2 hours before a meal, and 2 hours after a meal).
  Cycles 2 and beyond: Participants will take ASTX029 tablets by mouth every day (days 1-28) fasting, (2 hours before and 2 hours after a meal). You will also take ASTX727 tablets by mouth 1 time every day on days 1-5 of each cycle, fasting (2 hours before and 2 hours after a meal).
  Interventions: Drug: ASTX727; Drug: ASTX029-01

INTERVENTIONS:
Drug: ASTX727 — Given by PO
  Other Names: Inqovi
Drug: ASTX029-01 — Given by PO

SUMMARY:
To find the recommended dose of the study drugs ASTX727 and ASTX029 that can be given to patients with relapsed/refractory AML. The goal of Part 2 of the study is to learn if the dose of study drugs found in Part 1B can help to control AML.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the safety and recommended phase 2 dose (RP2D) of ASTX727 in combination with ASTX029 in patients with relapsed/refractory AML.

Secondary Objectives:

* To assess the CR+CRi+PR and MLFS rate within 6 cycles of treatment initiation of ASTX727 in combination with ASTX029 in patients with relapsed refractory AML.
* To determine the duration of response (DOR), event-free survival (EFS), overall survival (OS), minimal/measurable residual disease (MRD) status at response and best MRD response attained by flow-cytometry, 4- and 8-week mortality
* To investigate correlations of response to these combinations with a pre- therapy, on-therapy, and progression 81-gene panel of gene mutations in AML.

Exploratory Objectives:

* To investigate possible relationships between response and non-response to the combinations with myeloid mutation panel.
* To identify leukemic subpopulations and how their signaling state in disease relates to clinical outcomes by Flow cytometry or CyTOF (mass cytometry) on patients' bone marrow samples and/or peripheral blood baseline, on treatment, remission and relapse and potentially other time-points on study.
* To store and/or analyze surplus blood or tissue including bone marrow, if available, for potential future exploratory research into factors that may influence development of AML and/or response to the combination (where response is defined broadly to include efficacy, tolerability or safety).

ELIGIBILITY:
Inclusion Criteria:

* Phase 1B: Diagnosis of relapsed/refractory AML (excluding acute promyelocytic leukemia)
* Phase 2A: Diagnosis of relapsed/refractory AML (excluding acute promyelocytic leukemia) with MAPK pathway mutations e.g. N or KRAS, PTPN11, NF1 etc.

  1. Patients aged ≥18 years old with relapsed/refractory AML with MAPK pathway mutations e.g. N or KRAS, PTPN11, NF1 etc. are eligible if they are not eligible for potentially curative therapy such as more effective salvage therapy or hematopoietic stem cell transplantation or who refuse these options at the time of enrollment.
  2. Patient must be receiving protocol therapy as salvage 1 or 2.
* Phase 1B: Diagnosis of relapsed/refractory AML (excluding acute promyelocytic leukemia)
* Phase 2A: Diagnosis of relapsed/refractory AML (excluding acute promyelocytic leukemia) with MAPK pathway mutations e.g. N or KRAS, PTPN11, NF1 etc.

  1. Patients aged ≥18 years old with relapsed/refractory AML with MAPK pathway mutations e.g. N or KRAS, PTPN11, NF1 etc. are eligible if they are not eligible for potentially curative therapy such as more effective salvage therapy or hematopoietic stem cell transplantation or who refuse these options at the time of enrollment.
  2. Patient must be receiving protocol therapy as salvage 1 or 2.
  3. Patients aged ≥ 18 years old, with MDS or CMML treated with hypomethylating agent (HMA) therapies who progress to AML and have no available therapies or are not candidates for available therapies, will be eligible at the time of progression to AML.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
* Temporary prior measures such as apheresis while eligibility work-up is being performed are allowed and not counted as a prior salvage
* In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of protocol therapy will be at least 2 weeks or at least 5 half-lives (whichever is longer). The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator's brochures, or drug-administration manuals) and will be documented in the protocol eligibility document.
* The toxicity from prior therapy should have resolved to Grade ≤1, however alopecia and sensory neuropathy Grade ≤2 not constituting a safety risk based on investigators judgement is acceptable.
* The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following c: (1) intrathecal (IT) therapy for patients with controlled CNS leukemia at the discretion of the PI. (2) Use of 1-2 doses of cytarabine (up to 1.5 g/m2 each dose) for patients with rapidly proliferative disease is allowed up to 7 days before the start of study therapy (7 days washout). Since the anti-leukemia effect of HMA-therapies and kinase inhibitors may be delayed, use of hydroxyurea for patients with rapidly proliferative disease is allowed on study and before the start of study therapy and will not require a washout. These medications will be recorded in the case-report form. (Rationale: Patients with kinase mutations can have very proliferative disease and the combination can induce differentiation in patients as part of response)
* Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS disease is permitted. Patients with a known history of CNS disease must have been treated with CNS directed therapy, have at least 2 consecutive LPs with no evidence of CNS leukemia, and must be clinically stable for at least 4 weeks prior to enrollment and have no ongoing neurological symptoms that in the opinion of the treating physician are related to the CNS disease
* Serum biochemical values with the following limits:

  1. Patients must have adequate renal function as demonstrated by a creatinine clearance (CrCl) ≥ 50 mL/min calculated by either the Cockcroft-Gault formula, Modification of Diet in Renal Disease (MDRD) eGFR or measured by 24 hours' urine collection. For patients with BMI >23, Adjusted body weight and not Ideal Body Weight is the recommended parameter29, 30.
  2. Total bilirubin <1.5 x ULN unless considered due to Gilbert's syndrome
  3. Aspartate aminotransferase or alanine aminotransferase ≤2.0 x ULN (aspartate aminotransferase or alanine aminotransferase ≤3.0 x ULN if deemed related to leukemia by the treating physician)
* White blood cell count <15 x 109/L. Hydroxyurea may be used to reduce the WBC count to ≤ 15x109/L.
* Ability to understand and provide signed informed consent.
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment.
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 4 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment.

Exclusion Criteria:

* Patients with known allergy or hypersensitivity to ASTX727(Inqovi), ASTX029 or any of their components.
* Patients with known allergy or hypersensitivity to ASTX727(Inqovi), ASTX029 or any of their components.
* Patients with any other known concurrent severe and/or uncontrolled medical condition including but not limited to diabetes, cardiovascular disease including hypertension, renal disease, or active uncontrolled infection, which could compromise participation in the study.
* Patients on active antineoplastic or radiation therapy for a concurrent malignancy at the time of screening. Maintenance therapy, hormonal therapy, or steroid therapy for well-controlled malignancy is allowed.
* Prior organ transplantation including allogenic stem-cell transplantation within 3 months prior to planned enrollment, active graft versus host disease (GVHD) >Grade 1 or requiring transplant-related immunosuppression with the exception of low dose cyclosporine and tacrolimus.
* Prior treatment with an ERK inhibitor.
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including:

A) Presence of predisposing factors to RVO or CSR (eg, uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus) or b) Visible retinal pathology as assessed by ophthalmic examination at screening that is considered a risk factor for RVO or CSR such as:

* Evidence of optic disc cupping or
* Evidence of new visual field defects on automated perimetry or
* Intraocular pressure >21mmHg as measured by tonography.
* Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia.
* Patients with a known HIV infection that is not well controlled (i.e. any detectable circulating viral load) at the time of enrollment. No additional screening for HIV infection is needed.
* Patients with known positive hepatitis B or C infection by serology, with the exception of those with an undetectable viral load within 3 months (Hepatitis B or C testing is not required prior to study entry). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] may participate.
* Patients who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Patients who have had any major surgical procedure within 14 days of Day 1.
* Other severe acute or chronic medical conditions that is active and not well controlled including colitis, inflammatory bowel disease, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Active and uncontrolled disease (active infection requiring systemic therapy or fever likely secondary to infection within prior 48 hours): prophylactic antibiotics or prolonged course of IV antibiotics for controlled infection are allowed, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure NYHA class III/IV, clinically significant and uncontrolled arrhythmia) as judged by the treating physician.
* Patients unwilling or unable to comply with the protocol.
* Screening 12-lead ECG showing a Baseline average QT interval as corrected by Fridericia's formula (QTcF) >470 msec. Subjects with left or right bundle branch block, where QT cannot be accurately assessed, will be allowed into the study after assessment by institutional cardiologist
* Patients requiring strong CYP3A inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 [Time Frame: through study completion; an average of 1 year.]

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org